CLINICAL TRIAL: NCT01815905
Title: U-Health Service Using Mobile Device for Improvement of Post-Stroke Upper Limb Function and Aphasia
Brief Title: Effect of U-Health Service in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: KT Corporation (Industry)
Responsible Party: Principal Investigator, Nam-Jong Paik, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1206/160-005
Record Dates: First submitted 2013-03-11; First posted 2013-03-21 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional therapy (Active Comparator): Traditional rehabilitation therapy
  Interventions: Other: Traditional rehabilitation therapy
- Mobile program (Experimental): Mobile program for occupational and speech therapy
  Interventions: Other: Mobile program for occupational and speech therapy

INTERVENTIONS:
Other: Mobile program for occupational and speech therapy
  Arms: Mobile program
Other: Traditional rehabilitation therapy
  Arms: Traditional therapy

SUMMARY:
Provides mobile programs for occupational and speech therapy to patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* stroke confirmed by brain imaging study
* Impairment in upper extremity function or speech
* native speaker of Korean

Exclusion Criteria:

* previous history of aphasia
* psychiatric or psychotic problem
* severe cognitive dysfunction
* severe hearing or visual loss
* cannot sit with devices

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer upper extremity scale | 4weeks
  upper extremity function test
short form K-FAST (Korean version of Frenchay Aphasia Screening) | 4weeks
  speech function screening test

SECONDARY OUTCOMES:
Hand grip strength | 4weeks
  hand power measurement
K-WAB(Korean version-the Western Aphasia Battery) | 4weeks
  speech evaluation

OTHER OUTCOMES:
EuroQol(EQ-5D) | 4weeks
  measurement of health outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Bundang-gu, South Korea